CLINICAL TRIAL: NCT00134446
Title: A Prospective Double Blind Randomized Placebo Controlled Trial of Repetitive Transcranial Magnetic Stimulation for Posttraumatic Stress Disorder
Brief Title: Transcranial Magnetic Stimulation for Post-Traumatic Stress Disorder
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: White River Junction Veterans Affairs Medical Center (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WRJVAMC16744; Hitchcock Foundation
Record Dates: First submitted 2005-08-23; First posted 2005-08-24 (Estimated); Last update posted 2005-10-31 (Estimated); Status verified 2005-03

CONDITIONS: Post-Traumatic Stress Disorders
Keywords: post traumatic stress disorder; PTSD; trauma; transcranial magnetic stimulation; randomized clinical trial
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Wounds and Injuries | interventions — Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: transcranial magnetic stimulation

SUMMARY:
The purpose of this study is to determine if transcranial magnetic stimulation at 1 HZ to the right frontal cortex will decrease the symptoms of post-traumatic stress disorder (PTSD).

DETAILED DESCRIPTION:
Post-traumatic stress disorder (PTSD) is a psychiatric disorder that is common in the general population. PTSD symptoms include re-experiencing the traumatic event, avoidance of reminders of the trauma, and increased arousal. The primary treatments of PTSD are psychotherapy and antidepressant medications. While both are effective, many patients continue to have significant symptoms. Repetitive Transcranial Magnetic Stimulation (rTMS) is a new research and treatment modality that uses a small powerful electromagnet to directly stimulate the brain. This stimulation may increase or decrease brain activity. The treatments have been shown to be effective in other disorders such as depression. Initial treatment of patients with PTSD using rTMS has been hopeful. This study is the first randomized controlled trial to examine the efficacy of rTMS for PTSD.

This study would be the first randomized placebo controlled trial to examine the efficacy of Transcranial Magnetic Stimulation (rTMS) for PTSD. The primary hypothesis is that there will be significant improvement in the patients' PTSD symptoms from pre-treatment to post-treatment with rTMS. A secondary hypothesis is that the patients' co-morbid depressive symptoms will improve from pre-treatment to post-treatment. Forty subjects with PTSD will be recruited from the White River Junction VAMC. Patients will be randomly assigned to receive either active rTMS or sham rTMS. Patients, staff performing the treatments, and staff completing the assessments will all be blinded to active or sham treatment.

ELIGIBILITY:
Inclusion Criteria:

* PTSD diagnosis on standardized assessment
* Medically stable
* Eligible veteran of United States (US) military

Exclusion Criteria:

* Active substance abuse
* History of seizures
* Metal in head or neck

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2004-03

PRIMARY OUTCOMES:
Clinician-Administered PTSD Scale (CAPS)

SECONDARY OUTCOMES:
PTSD Clinician Checklist (PCL)
Beck Depression Inventory (BDI)
State-Trait Anxiety Inventory (STAI)
Side Effect Checklist
Brief Cognitive Examination

CONTACTS AND LOCATIONS:
Overall Officials: Bradley V Watts, MD, Principal Investigator — White River Junction Veterans Affairs Medical Center
Locations (1):
- White River Junction VAMC, White River Junction, Vermont, United States